CLINICAL TRIAL: NCT05901571
Title: Acupuncture and Escitalopram for Treating Major Depression Clinical Study (AE-TMDCS): Study Design of a Randomized Controlled Trial
Brief Title: Acupuncture and Escitalopram for Treating Major Depression Clinical Study
Acronym: AE-TMDCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 7th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PWRl2021-05; 21Y11921000 (Other Grant/Funding Number: Shanghai science and techonology committe); 21ZR1449300 (Other Grant/Funding Number: Natural Science Foundation of Shanghai)
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acupuncture Therapy; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sham-acupuncture/placebo-pill (Sham Comparator): sham-acupuncture protocol plus escitalopram placebo
  Interventions: Other: sham-acupuncure; Other: escitalopram placebo
- sham-acupuncture/escitalopram (Active Comparator): sham-acupuncture protocol plus escitalopram
  Interventions: Other: escitalopram; Other: sham-acupuncure
- active acupuncture/placebo-pill (Active Comparator): acupuncture protocol plus escitalopram placebo
  Interventions: Other: acupuncture; Other: escitalopram placebo
- active acupuncture/escitalopram (Experimental): acupuncture protocol plus escitalopram
  Interventions: Other: acupuncture; Other: escitalopram

INTERVENTIONS:
Other: acupuncture — The acupuncture group will receive treatment with needles inserted at the specified acupoints. Selected by acupuncture experts, these acupoints include SP4 (Gongsun) , PC6 (Neiguan) , PC5 (Jianshi) and LV 3 (Taichong) bilaterally. All acupoints are localized according to the WHO Standard Acupuncture Locations.After needle insertion, the acupuncture needles will be manipulated using either the twirling-rotating or lifting-thrusting methods to achieve the "De Qi" sensation.
  Other Names: active acupuncture
  Arms: active acupuncture/escitalopram; active acupuncture/placebo-pill
Other: escitalopram — Patients will receive 10 mg/day of escitalopram for the first 3 weeks and 20mg/day for the remaining 7 weeks.
  Arms: active acupuncture/escitalopram; sham-acupuncture/escitalopram
Other: sham-acupuncure — In the sham acupuncture group, superficial skin penetration (2 to 3 mm in depth) at nonacupoints will be done without De Qi manipulations. Nonacupoints are away from conventional acupoints or meridians. The choice of sham acupuncture points, which are points located in an emplacement different than the meridian points. The sham acupoints are not standard acupoints and will be about 1cun ( ≈20 mm) lateral from the real acupoints in the experimental group.
  Arms: sham-acupuncture/escitalopram; sham-acupuncture/placebo-pill
Other: escitalopram placebo — Patients will receive 10 mg/day of escitalopram placebo for the first 3 weeks and 20mg/day for the remaining 7 weeks.
  Arms: active acupuncture/placebo-pill; sham-acupuncture/placebo-pill

SUMMARY:
We will be able to investigate in a sample of patients free of antidepressants whether acupuncture is more effective than placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, 2 by 2 factorial clinical trial for Major depression.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years of age with no gender-based restriction.
2. Fulfilling the diagnostic criteria of DSM-5 for major depressive disorder.
3. A Hamilton Rating Scale for Depression (HDRS-17) score ≥ 17
4. Ability to read and understand Mandarin Chinese, at least nine years of education, and willingness to adhere to the study protocol.
5. The absence of acupuncture treatment within at least 1 year.
6. Willingness to participate in the trial and provide written informed consent for the clinical trial.

Exclusion Criteria:

1. Lifetime or current neuropsychiatric conditions, such as bipolar disorder, schizophrenia, substance dependence or abuse, dementia, brain injury, epilepsy and so forth.
2. High suicide risk or presenting with suicidal ideation (a score of more than 2 points on the Suicide question of the HDRS-17) at the time of entry.
3. Medicated with antidepressant at the start of the trial or history of treatment failure to escitalopram.
4. Pregnancy or breastfeeding.
5. Subjects who have acute inflammation at the planned acupuncture site on the body or any other contraindication to acupuncture.
6. Candidates afraid of needles in general and reluctant to receive acupuncture in particular
7. Known or suspected clinically unstable systemic medical disorder (including cancer, organ failure, or severe diseases of the cardiovascular, severe hepatic or renal insufficiency).
8. Previous participation in other acupuncture trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
HDRS-17 score | from baseline to 10 weeks
  the change in the HDRS-17 score

SECONDARY OUTCOMES:
Beck depression inventory score | from baseline to 10 weeks
  the change in the Beck depression inventory score
The CGI(Clinical Global Impression) | from baseline to 10 weeks
  the change in the CGI
The GAD-7(General Anxiety Disorder) | from baseline to 10 weeks
  the change in the GAD-7
The Mini-Mental State Examination (MMSE) | from baseline to 10 weeks
  the change in the MMSE

OTHER OUTCOMES:
BDNF | at baseline and 10 week
  serum BDNF level
IL18/IL-1β | at baseline and 10 week
  serum IL18/IL-1β level
fMRI | at baseline and 10 week
  functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Zhenxiang Han, Dr, Principal Investigator — Shanghai Seventh People's Hospital, Shanghai University of TCM
Locations (3):
- China (3):
  - Jianhua Chen, Shanghai, Shanghai Municipality
  - Zhenxiang Han, Shanghai, Shanghai Municipality
  - Zouqing Huang, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
The paper will be published.
Supporting Information: Study Protocol, SAP
Access Criteria: ResMan IPD
URL: http://www.medresman.org.cn

REFERENCES:
- [Derived] Yang K, Tiwari S, Liu D, Xu Q, Qi L, Zhu Y, Jiang L, Zouqin H, Wong J, Chen J, Han Z. Acupuncture and Escitalopram for Treating Major Depression Clinical Study (AE-TMDCS): protocol for a factorial randomised controlled trial. BMJ Open. 2024 Sep 10;14(9):e091214. doi: 10.1136/bmjopen-2024-091214. PMID 39260834